CLINICAL TRIAL: NCT03387423
Title: ESCALATE-RA A NON-INTERVENTIONAL STUDY OF CRITICAL FACTORS FOR ESCALATING DRUG TREATMENT IN PATIENTS TREATED WITH TOFACITINIB FOR MODERATE TO SEVERE ACTIVE RHEUMATOID ARTHRITIS
Brief Title: Observational Study to Determine How Physicians Make Treatment Decisions in Patients Treated With Tofacitinib for Moderate to Severe Active Rheumatoid Arthritis
Acronym: ESCALATE-RA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921302; ESCALATE-RA (Other: Alias Study Number)
Record Dates: First submitted 2017-12-07; First posted 2018-01-02 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Tofacitinib — Patients who are started on Tofacitinib treatment according to the drug label

SUMMARY:
This non-interventional study aims to identify key factors that are driving treatment decisions by rheumatologists in the treatment of rheumatoid arthritis (RA) patients starting treatment with Tofacitinib in a real world setting.

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥ 18 years

Confirmed Diagnosis of Rheumatoid Arthritis by rheumatologist

Patient is eligible for Tofacitinib treatment according to Summary of Product Characteristics (SmPC)

Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

Contraindications according to Xeljanz® SmPC

Receipt of any investigational drug within 3 months before study inclusion

Patients who have received any previous treatment with Tofacitinib or other JAK inhibitors

Patients who are investigational site staff members or patients who are Pfizer employees directly involved in the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with confirmed diagnosis of rheumatoid arthritis who are eligible for treatment with Tofacitinb according to Summary of Product Characteristics (SmPC)
Sampling Method: Non-Probability Sample
Enrollment: 1459 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (91):
- Germany (91):
  - Private Praxis, Düsseldorf, North Rhine-Westphalia
  - Private Practice, Zschopau, Saxony
  - Private Practice Kupka, Altenburg
  - Private Practise Boehm, Altenholz
  - Private Practice Marycz, Amberg
  - Private Practice Fuchs, Augsburg
  - private practise Gause, Bad Bramstedt
  - ACURA Kliniken Rheinland-Pfalz AG, Bad Kreuznach
  - MFZ Medizinisches Forschungszentrum Weserbergland, Bad Pyrmont
  - Private Practice Manger, Bamberg
  - Private Practice Ochs, Bayreuth
  - Private Practice Schmitt-Haendle, Bayreuth
  - Private Practice, Bayreuth
  - Ambulantes Gesundheitszentrum der Charité, Berlin
  - Private Practice Bozorg, Berlin
  - Private Practice Brandt-Juergens, Berlin
  - Privat Practice Remstedt, Berlin
  - private practise Herzberg, Berlin
  - Private Practice Seifert, Berlin
  - Private Practice Zinke, Berlin
  - Private Practice Thiele, Berlin
  - Immanuel Klinikum Bernau, Bernau
  - Private Practise, Braunschweig
  - MED Bayern OST GmbH, Burghausen
  - Private Practice Lorenz, Chemnitz
  - Private Practice Baerlecken, Cologne
  - Private Practice Kirrstetter, Deggendorf
  - Kreiskranenhaus Demmin GmbH, Demmin
  - Private Practice Menne, Dortmund
  - Private Practice Luethke, Dresden
  - Private Practice Fischer, Dresden
  - private practise Pech, Eberswalde
  - Private Practice Steinmueller, Ehringshausen
  - Asklepios MVZ Nord SH GmbH, c/o AK St. Georg, Elmshorn
  - Private Practice Kaestner, Erfurt
  - Private Practice Koch, Erfurt
  - Private Practice Haeckel, Frankenberg
  - Private Practice Mueller, Freiberg
  - SRH Krankenhaus Waltershausen-Friedrichroda GmbH, Friedrichroda
  - Private Practice Abahji, Germering
  - Private Practice Sensse, Gifhorn
  - Private Practice Holst, Glaisin
  - Private Practice Zeh, Göppingen
  - Private Practice Semmler, Güstrow
  - private practise Kühne, Haldensleben I
  - Private Practice Liebhaber, Halle
  - Private Practice Dahmen, Hamburg
  - private practise Aries, Hamburg
  - Private Practice Stille, Hanover
  - private practise Heilig, Heidelberg
  - private practise Wernicke, Hohen Neuendorf
  - Private Practice Kremers, Jülich
  - Medius Kliniken gGmbH, Kirchheim unter Teck
  - Kreiskrankenhaus Langenau, Langenau
  - Private Practice Hamann, Leipzig
  - Private Practice Schwarze, Leipzig
  - Private Practice Kudela, Magdeburg
  - private practise Sieburg, Magdeburg
  - Private Practice Rossbach, Mansfeld
  - Private Practice Harmuth, Marktredwitz
  - Private Practice Worsch, Mühlhausen
  - Private Practice Krueger, München
  - Private Practice Raub, Münster
  - Praxis Dr.med. Holger Krauel Facharzt für Innere Medizin und Rheumatologie, Naumburg
  - Private Practice Berger, Naunhof
  - Private Practise, Neubrandenburg
  - Private Practice Volberg, Neuss
  - MCN Medic Center Nuernberg GmbH, Nuremberg
  - Private Practice Goettl, Passau
  - Private Practice Graessler, Pirna
  - Private Practice Baumann, Plauen
  - Knappschaftsklinikum Soor, Klinik fuer Rheumatologie und Klinische Immunologie, Püttlingen
  - Private Practice Wassenberg, Koehler, Weier, Ratingen
  - Private Practice Richter, Rostock
  - private practise Biewer, Saarbrücken
  - MVZ Dialysezentrum Schweinfurt, Schweinfurt
  - Private Practice Moebius, Schwerin
  - Private Practice, Schwerin
  - private practise Ständer, Schwerin
  - Private Practice Melzer, Seesen
  - MVZ Klinikum Straubing, Straubing
  - Private Practice, Templin
  - Private Practice Pyra, Torgelow
  - Private Practice Haas, Tübingen
  - Klinik an der Weissenburg GmbH, Uhlstaedt-Kirchhasel
  - Private Practice Rinaldi, Ulm
  - Private Practice Woerth, Wiesbaden
  - Klinikverbund St. Antonius und St. Josef GmbH, Wuppertal
  - Rheuma Praxis Barmen Dres. med. Demirel / Hruschka, Wuppertal
  - Private Practice Fricke-Wagner, Zwickau
  - Private Practice Alliger, Zwiesel

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 1518 participants were screened in this observational study, out of which 1459 eligible participants were enrolled and 59 we excluded. Out of these 59 participants, 30 participants were excluded due to retrospective screening failure and data review meeting decision as the type of therapy (monotherapy or combination therapy) was not defined and 29 participants were not eligible as their treatment with Tofacitinib was not started.
Pre-assignment Details: Data from German participants with rheumatoid arthritis (RA) who initiated treatment with Tofacitinib or switched to other therapies from initial tofacitinib therapy in real world setting were observed for 24 months in this non-interventional observational study.
Groups:
- Tofacitinib Monotherapy: Participants who were on tofacitinib monotherapy treatment throughout the study as part of their routine clinical treatment were followed up for 24 months from the date of first tofacitinib prescription. Treatment dose and frequency of follow-up were decided by the treating physician.
- Tofacitinib+Methotrexate (MTX) Combination Therapy: Participants who were on combination therapy of tofacitinib with Methotrexate (MTX) throughout the study as part of their routine clinical treatment were followed up for 24 months from the date of first tofacitinib prescription. Treatment dose and frequency of follow-up were decided by the treating physician.
- Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy: Participants who were on tofacitinib monotherapy and then switched to tofacitinib +MTX combination therapy as part of their routine clinical treatment were followed up for 24 months from the date of first tofacitinib prescription. Treatment dose and frequency of follow-up were decided by the treating physician.
- Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy: Participants who were on combination therapy of tofacitinib+MTX and then switched to tofacitinib monotherapy as part of their routine clinical treatment were followed up for 24 months from the date of first tofacitinib prescription. Treatment dose and frequency of follow-up were decided by the treating physician.
Period: Overall Study
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Started | 779 | 440 | 111 | 129
Completed | 521 | 304 | 90 | 105
Not Completed | 258 | 136 | 21 | 24
Not completed — Lost to Follow-up | 16 | 12 | 1 | 0
Not completed — Other | 0 | 3 | 0 | 0
Not completed — Administrative Reason | 166 | 89 | 17 | 19
Not completed — Revocation Consent | 76 | 32 | 3 | 5

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy | Total
Number analyzed (Participants) | 779 | 440 | 111 | 129 | 1459
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 90 | 43 | 13 | 22 | 168
  45-64 years | 389 | 287 | 75 | 61 | 812
  More than or equal to (>=) 65 years | 300 | 110 | 23 | 46 | 479
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 627 | 307 | 90 | 91 | 1115
  Male | 152 | 133 | 21 | 38 | 344
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Escalations
Description: Treatment escalations was defined as participants who switched to another disease modifying antirheumatic drug (DMARD) or combination of DMARDs when compared to the last visit. The following three types of escalations were reported: treatment termination, treatment step-up/switch and treatment step-down. Treatment termination was defined as the termination of a DMARD (or multiple when on combination therapy) without starting a new DMARD therapy. Treatment step-up/switch was defined as an increase from the current treatment regime towards e.g.a combination of DMARDs and treatment step-down, was defined as de-escalation from the current treatment regime, example (e.g.) from combination therapy to monotherapy. One participant can fall into more than 1 type of escalation.
Time Frame: From date of first prescription of tofacitinib up to 24 Months
Population: Full analysis set (FAS) included all participants who received at least 1 dose of tofacitinib and had at least 1 set of post-baseline measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Step-up/switch | 249 | 130 | 101 | 48
  Step-down | 29 | 51 | 39 | 91
  Treatment termination | 109 | 2 | 7 | 26
  Any escalation | 341 | 156 | 111 | 123

2. Primary Outcome: Time to Treatment Escalation
Description: Time to treatment escalation was defined as time in days from escalation visit date to next escalation visit date. The following three types of escalations were reported: treatment termination, treatment step-up/switch and treatment step-down. Treatment termination was defined as the termination of a DMARD (or multiple when on combination therapy) without starting a new DMARD therapy. Treatment step-up/switch was defined as an increase from the current treatment regime (monotherapy) towards a combination of DMARDs and treatment step-down, was defined as de-escalation from the current treatment regime, e.g. from combination therapy to monotherapy. Number of participants with total number of each type of treatment escalations during the study (step-up/switch, step-down, treatment termination along with all escalations) are reported in this outcome measure.
Time Frame: From date of first prescription of tofacitinib up to 24 Months
Population: FAS included all participants who received at least 1 dose of tofacitinib and had at least 1 set of post-baseline measurements. Here" Number analyzed" signifies participants evaluable for specific rows.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 341 | 156 | 111 | 123
Days
  All Escalations: 1 Treatment escalation | 288.21 (210.01) | 278.47 (188.96) | 221.95 (154.99) | 308.11 (190.70)
  All Escalations: 2 Treatment escalation: number analyzed (Participants) | 96 | 53 | 66 | 45
  All Escalations: 2 Treatment escalation | 240.39 (162.67) | 219.47 (152.66) | 234.58 (154.80) | 239.20 (166.14)
  All Escalations: 3 Treatment escalation: number analyzed (Participants) | 34 | 13 | 32 | 17
  All Escalations: 3 Treatment escalation | 175.56 (117.36) | 258.92 (153.07) | 216.84 (137.04) | 193.35 (126.70)
  All Escalations: 4 Treatment escalation: number analyzed (Participants) | 7 | 0 | 8 | 3
  All Escalations: 4 Treatment escalation | 211.43 (133.53) |  | 202.88 (101.76) | 186.33 (60.67)
  All Escalations: 5 Treatment escalation: number analyzed (Participants) | 1 | 0 | 3 | 1
  All Escalations: 5 Treatment escalation | 92.00 |  | 94.00 (4.36) | 160.00
  All Escalations: 6 Treatment escalation: number analyzed (Participants) | 0 | 0 | 0 | 1
  All Escalations: 6 Treatment escalation |  |  |  | 106.00
  Step up/switch: 1 Treatment escalation: number analyzed (Participants) | 249 | 130 | 101 | 48
  Step up/switch: 1 Treatment escalation | 303.14 (214.45) | 286.58 (196.41) | 240.05 (169.23) | 273.15 (164.79)
  Step up/switch: 2 Treatment escalation: number analyzed (Participants) | 69 | 30 | 51 | 23
  Step up/switch: 2 Treatment escalation | 236.51 (170.99) | 242.07 (156.23) | 248.78 (169.24) | 258.74 (191.11)
  Step up/switch: 3 Treatment escalation: number analyzed (Participants) | 24 | 7 | 17 | 6
  Step up/switch: 3 Treatment escalation | 196.88 (129.53) | 194.71 (116.10) | 196.24 (109.94) | 188.33 (119.09)
  Step up/switch: 4 Treatment escalation: number analyzed (Participants) | 4 | 0 | 5 | 2
  Step up/switch: 4 Treatment escalation | 208.25 (172.07) |  | 185.40 (108.18) | 231.50 (129.40)
  Step up/switch: 5 Treatment escalation: number analyzed (Participants) | 0 | 0 | 2 | 0
  Step up/switch: 5 Treatment escalation |  |  | 95.50 (4.95) |
  Step down: 1 Treatment escalation: number analyzed (Participants) | 29 | 51 | 39 | 91
  Step down: 1 Treatment escalation | 304.55 (222.48) | 381.24 (212.79) | 392.46 (238.26) | 362.63 (201.10)
  Step down: 2 Treatment escalation: number analyzed (Participants) | 0 | 2 | 0 | 0
  Step down: 2 Treatment escalation |  | 480.00 (5.66) |  |
  Treatment termination: 1 Treatment escalation: number analyzed (Participants) | 104 | 2 | 5 | 20
  Treatment termination: 1 Treatment escalation | 336.52 (228.53) | 137.50 (64.35) | 520.80 (264.57) | 485.70 (246.06)

3. Secondary Outcome: Time to First Step Up Treatment Escalation
Description: Time to first step-up treatment escalation was defined for participants who experienced a treatment step-up and was measured as date of first treatment step up escalation minus (-) date of first prescription of tofacitinib. Treatment step-up was defined as an increase from the current treatment regime (monotherapy) towards a combination of DMARDs.
Time Frame: From date of first tofacitinib prescription up to date of first step-up treatment escalation (maximum up to 24 months)
Population: FAS included all participants who received at least 1 dose of tofacitinib and had at least 1 set of post-baseline measurements.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Days | 611.33 (10.27) | 599.17 (12.38) | 268.07 (19.86) | 555.69 (21.68)

4. Secondary Outcome: Number of Participants Achieving Low Disease Activity (LDA) as Assessed by Simplified Disease Activity Index (SDAI) at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: SDAI was calculated using the following formula: SDAI = Tender Joint Count (TJC) (using 28 joints) + Swollen Joint Count (SJC) (using 28 joints) + Patient Global Assessment of Arthritis (PtGA) (0-10 centimetre [cm] scale) + Physician's Global Assessment of Arthritis (PhGA) (0-10 cm scale) + C-reactive protein (CRP) (milligram per decilitre [mg/dL]). TJC28 joints included shoulders, elbows, wrists, metacarpophalangeal (MCP) and proximal interphalangeal (PIP) joints, and knees whereas SJC28 included shoulders, elbows, wrists, MCP, PIP and knees (excluding artificial joints). PtGA and PhGA both were assessed on 0-10 cm visual analogue scale (VAS) scale (0 cm [very well] to 10 cm [worst], where higher scores indicated greater affliction due to disease activity). SDAI total score ranged from 0 to 86, where higher scores indicated higher disease activity. SDAI score of less than or equal to (<=11) indicates LDA.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: Secondary FAS (SFAS): all participants who received at least 1 dose of tofacitinib, had >=1 set of post-baseline values & whose data was collected while taking tofacitinib. A participant was considered on tofacitinib at a given timepoint if tofacitinib was not terminated/paused at time of the visit/event. "Number Analyzed"=participants evaluable for specified rows. All participants reported under "Number of Participants Analyzed' contributed data but may not have evaluable data for every row.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Month 3: number analyzed (Participants) | 479 | 278 | 69 | 94
  Month 3 | 281 | 164 | 31 | 63
  Month 6: number analyzed (Participants) | 383 | 229 | 51 | 78
  Month 6 | 256 | 127 | 22 | 56
  Month 9: number analyzed (Participants) | 328 | 203 | 38 | 67
  Month 9 | 225 | 134 | 16 | 48
  Month 12: number analyzed (Participants) | 303 | 191 | 29 | 61
  Month 12 | 221 | 131 | 17 | 45
  Month 15: number analyzed (Participants) | 262 | 162 | 15 | 56
  Month 15 | 197 | 109 | 8 | 42
  Month 18: number analyzed (Participants) | 237 | 159 | 15 | 53
  Month 18 | 159 | 114 | 9 | 39
  Month 21: number analyzed (Participants) | 228 | 144 | 14 | 49
  Month 21 | 166 | 99 | 8 | 37
  Month 24: number analyzed (Participants) | 209 | 149 | 12 | 49
  Month 24 | 149 | 111 | 6 | 41

5. Secondary Outcome: Number of Participants Achieving LDA as Assessed by Clinical Disease Activity Index (CDAI) at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: CDAI was calculated using the following formula: CDAI = (28TJC) + (28SJC) + (PhyGA in cm) + (PtGA in cm). TJC28 joints included shoulders, elbows, wrists, MCP and proximal PIP joints, and knees whereas SJC28 included shoulders, elbows, wrists, MCP, PIP and knees (excluding artificial joints). PtGA and PhGA both were assessed on 0-10 cm VAS scale (0 cm [very well] to 10 cm [worst], where higher scores indicated greater affliction due to disease activity). CDAI total score ranged from 0 to 76, where higher scores indicated higher disease activity. CDAI score of <= 10 indicates LDA.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: SFAS: all participants who received at least 1 dose of tofacitinib, had >=1 set of post-baseline values & whose data was collected while taking tofacitinib. A participant was considered on tofacitinib at a given timepoint if tofacitinib was not terminated/paused at time of the visit/event. "Number Analyzed"=participants evaluable for specified rows. All participants reported under "Number of Participants Analyzed' contributed data but may not have evaluable data for every row.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Month 3: number analyzed (Participants) | 593 | 345 | 88 | 108
  Month 3 | 348 | 197 | 40 | 71
  Month 6: number analyzed (Participants) | 486 | 281 | 61 | 94
  Month 6 | 315 | 162 | 28 | 65
  Month 9: number analyzed (Participants) | 416 | 254 | 50 | 80
  Month 9 | 293 | 172 | 25 | 57
  Month 12: number analyzed (Participants) | 375 | 223 | 38 | 75
  Month 12 | 266 | 154 | 23 | 56
  Month 15: number analyzed (Participants) | 344 | 205 | 22 | 65
  Month 15 | 254 | 144 | 13 | 49
  Month 18: number analyzed (Participants) | 311 | 191 | 20 | 62
  Month 18 | 205 | 141 | 13 | 46
  Month 21: number analyzed (Participants) | 292 | 178 | 18 | 57
  Month 21 | 204 | 130 | 11 | 45
  Month 24: number analyzed (Participants) | 272 | 178 | 16 | 61
  Month 24 | 199 | 135 | 9 | 51

6. Secondary Outcome: Number of Participants Achieving LDA Based on Disease Activity Score (DAS28-4) Erythrocyte Sedimentation Rate (ESR) at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated using the following formula: 0.56* square root of (TJC28) + 0.28* square root of (SJC28) + 0.70* natural log (ln) (ESR in [millimeter per hour [mm/ hour]) + 0.014*(PtGA in cm). PtGA was assessed on 0-10 cm VAS scale (scores ranging from 0 cm [very well] to 10 cm [worst]), where higher scores indicated greater affliction due to disease activity). Total DAS28-4 (ESR) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 ESR <= 3.2 indicates LDA.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Month 3: number analyzed (Participants) | 467 | 287 | 67 | 88
  Month 3 | 253 | 155 | 32 | 57
  Month 6: number analyzed (Participants) | 390 | 233 | 53 | 72
  Month 6 | 224 | 131 | 21 | 49
  Month 9: number analyzed (Participants) | 336 | 209 | 39 | 63
  Month 9 | 204 | 116 | 15 | 42
  Month 12: number analyzed (Participants) | 310 | 204 | 28 | 58
  Month 12 | 200 | 131 | 16 | 39
  Month 15: number analyzed (Participants) | 271 | 174 | 19 | 52
  Month 15 | 157 | 108 | 12 | 37
  Month 18: number analyzed (Participants) | 262 | 165 | 18 | 51
  Month 18 | 161 | 107 | 11 | 32
  Month 21: number analyzed (Participants) | 244 | 254 | 14 | 48
  Month 21 | 147 | 103 | 7 | 32
  Month 24: number analyzed (Participants) | 215 | 153 | 13 | 47
  Month 24 | 138 | 101 | 8 | 32

7. Secondary Outcome: Number of Participants Achieving LDA as Based on DAS28-4 C-Reactive Protein (CRP) at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (CRP) was calculated using the following formula: 0.56* square root of (TJC28) + 0.28* square root of (SJC28) + 0.36*ln (CRP in mg/l +1) + 0.014*(PtGA in mm)+ 0.96. PtGA was assessed on 0-10 cm VAS scale (scores ranging from 0 cm [very well] to 10 cm [worst]), where higher scores indicated greater affliction due to disease activity). Total DAS28-4 (CRP) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 CRP <= 3.2 indicates LDA.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Month 3: number analyzed (Participants) | 480 | 280 | 69 | 94
  Month 3 | 308 | 175 | 38 | 65
  Month 6: number analyzed (Participants) | 385 | 231 | 51 | 78
  Month 6 | 280 | 136 | 24 | 60
  Month 9: number analyzed (Participants) | 330 | 204 | 38 | 67
  Month 9 | 250 | 144 | 19 | 54
  Month 12: number analyzed (Participants) | 305 | 192 | 29 | 61
  Month 12 | 234 | 137 | 17 | 47
  Month 15: number analyzed (Participants) | 263 | 164 | 15 | 56
  Month 15 | 202 | 115 | 10 | 42
  Month 18: number analyzed (Participants) | 239 | 159 | 15 | 54
  Month 18 | 172 | 117 | 10 | 42
  Month 21: number analyzed (Participants) | 228 | 144 | 14 | 49
  Month 21 | 174 | 110 | 8 | 38
  Month 24: number analyzed (Participants) | 210 | 149 | 12 | 49
  Month 24 | 156 | 117 | 6 | 41

8. Secondary Outcome: Number of Participants Achieving Remission as Assessed by American College of Rheumatology (ACR)-EULAR Boolean Remission Criteria at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: ACR-EULAR Boolean remission criteria was defined as when participant had ACR remission =1 if; TJC28 <=1, SJC28 <=1, CRP <=1mg/dL and PtGA <= 2 cm on a 0 to 10 cm scale, where higher values indicate greater affection due to disease activity.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Month 3: number analyzed (Participants) | 480 | 280 | 69 | 94
  Month 3 | 21 | 15 | 1 | 8
  Month 6: number analyzed (Participants) | 385 | 231 | 51 | 78
  Month 6 | 22 | 13 | 0 | 6
  Month 9: number analyzed (Participants) | 330 | 204 | 38 | 67
  Month 9 | 25 | 9 | 1 | 0
  Month 12: number analyzed (Participants) | 305 | 192 | 29 | 61
  Month 12 | 28 | 12 | 1 | 2
  Month 15: number analyzed (Participants) | 263 | 264 | 15 | 56
  Month 15 | 11 | 5 | 1 | 4
  Month 18: number analyzed (Participants) | 239 | 159 | 15 | 54
  Month 18 | 11 | 11 | 0 | 2
  Month 21: number analyzed (Participants) | 228 | 144 | 14 | 49
  Month 21 | 13 | 12 | 1 | 2
  Month 24: number analyzed (Participants) | 210 | 149 | 12 | 49
  Month 24 | 11 | 7 | 0 | 4

9. Secondary Outcome: Number of Participants Achieving Remission as Assessed by SDAI at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: SDAI was calculated using the following formula: SDAI = (TJC28) + (SJC28) + (PtGA in cm) + (PhGA in cm) + (CRP in mg/dL). TJC28 joints included shoulders, elbows, wrists, MCP and PIP joints, and knees whereas SJC28 included shoulders, elbows, wrists, MCP, PIP and knees (excluding artificial joints). PtGA and PhGA both were assessed on 0-10 cm VAS scale (0 cm [very well] to 10 cm [worst], where higher scores indicated greater affliction due to disease activity). SDAI total score ranged from 0 to 86, where higher scores indicated higher disease activity. SDAI score of <=3.3 indicates remission.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Month 3: number analyzed (Participants) | 479 | 278 | 69 | 94
  Month 3 | 72 | 47 | 4 | 21
  Month 6: number analyzed (Participants) | 383 | 229 | 51 | 78
  Month 6 | 71 | 40 | 2 | 22
  Month 9: number analyzed (Participants) | 328 | 203 | 38 | 67
  Month 9 | 73 | 43 | 2 | 15
  Month 12: number analyzed (Participants) | 303 | 191 | 29 | 61
  Month 12 | 78 | 40 | 4 | 16
  Month 15: number analyzed (Participants) | 262 | 162 | 15 | 66
  Month 15 | 48 | 34 | 3 | 15
  Month 18: number analyzed (Participants) | 237 | 159 | 15 | 53
  Month 18 | 48 | 39 | 2 | 15
  Month 21: number analyzed (Participants) | 228 | 144 | 14 | 49
  Month 21 | 51 | 34 | 4 | 17
  Month 24: number analyzed (Participants) | 209 | 149 | 12 | 49
  Month 24 | 46 | 38 | 2 | 21

10. Secondary Outcome: Number of Participants Achieving Remission as Assessed by CDAI at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: CDAI was calculated using the following formula: CDAI = (28TJC) + (28SJC) + (PhyGA in cm) + (PtGA in cm). TJC28 joints included shoulders, elbows, wrists, MCP and proximal PIP joints, and knees whereas SJC28 included shoulders, elbows, wrists, MCP, PIP and knees (excluding artificial joints). PtGA and PhGA both were assessed on 0-10 cm VAS scale (0 cm [very well] to 10 cm [worst], where higher scores indicated greater affliction due to disease activity). CDAI total score ranged from 0 to 76, where higher scores indicated higher disease activity. CDAI score of <=2.8 indicates remission.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Month 3: number analyzed (Participants) | 593 | 345 | 88 | 108
  Month 3 | 94 | 65 | 8 | 28
  Month 6: number analyzed (Participants) | 486 | 281 | 61 | 94
  Month 6 | 96 | 61 | 5 | 27
  Month 9: number analyzed (Participants) | 416 | 254 | 50 | 80
  Month 9 | 84 | 59 | 5 | 19
  Month 12: number analyzed (Participants) | 375 | 223 | 38 | 75
  Month 12 | 98 | 51 | 6 | 18
  Month 15: number analyzed (Participants) | 344 | 205 | 22 | 65
  Month 15 | 67 | 55 | 6 | 17
  Month 18: number analyzed (Participants) | 311 | 191 | 20 | 62
  Month 18 | 68 | 51 | 4 | 20
  Month 21: number analyzed (Participants) | 292 | 178 | 18 | 57
  Month 21 | 68 | 49 | 8 | 23
  Month 24: number analyzed (Participants) | 272 | 178 | 16 | 61
  Month 24 | 69 | 53 | 3 | 26

11. Secondary Outcome: Number of Participants Achieving Remission as Assessed by DAS-28 ESR at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated using the following formula: 0.56*square root of (TJC28) + 0.28*square root of (SJC28) + 0.70*In (ESR in mm/ hour) + 0.014*PtGA in cm. PtGA was assessed on 0-10 cm VAS scale (scores ranging from 0 cm [very well] to 10 cm [worst]), where higher scores indicated greater affliction due to disease activity). Total DAS28-4 (ESR) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 ESR score of <2.6 indicates remission.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Month 3: number analyzed (Participants) | 467 | 287 | 67 | 88
  Month 3 | 162 | 101 | 17 | 45
  Month 6: number analyzed (Participants) | 390 | 233 | 53 | 72
  Month 6 | 143 | 97 | 9 | 32
  Month 9: number analyzed (Participants) | 336 | 209 | 39 | 63
  Month 9 | 139 | 80 | 9 | 27
  Month 12: number analyzed (Participants) | 310 | 204 | 28 | 58
  Month 12 | 136 | 90 | 6 | 22
  Month 15: number analyzed (Participants) | 271 | 174 | 19 | 52
  Month 15 | 100 | 76 | 5 | 25
  Month 18: number analyzed (Participants) | 262 | 165 | 18 | 51
  Month 18 | 102 | 76 | 8 | 23
  Month 21: number analyzed (Participants) | 244 | 154 | 14 | 48
  Month 21 | 92 | 65 | 6 | 22
  Month 24: number analyzed (Participants) | 215 | 153 | 13 | 47
  Month 24 | 80 | 68 | 5 | 26

12. Secondary Outcome: Number of Participants Achieving Remission as Assessed by DAS28-4 CRP at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (CRP) was calculated using the following formula: 0.56*square root of (TJC28) + 0.28*square root of (SJC28) + 0.36*ln (CRP in mg/l +1) + 0.014*(PtGA in cm)+ 0.96. PtGA was assessed on 0-10 cm VAS scale (scores ranging from 0 cm [very well] to 10 cm [worst]), where higher scores indicated greater affliction due to disease activity). Total DAS28-4 (CRP) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 CRP score of <2.6 indicates remission.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Month 3: number analyzed (Participants) | 480 | 280 | 69 | 94
  Month 3 | 238 | 125 | 27 | 55
  Month 6: number analyzed (Participants) | 385 | 231 | 51 | 78
  Month 6 | 208 | 104 | 19 | 52
  Month 9: number analyzed (Participants) | 330 | 204 | 38 | 67
  Month 9 | 199 | 103 | 14 | 41
  Month 12: number analyzed (Participants) | 305 | 192 | 29 | 61
  Month 12 | 196 | 110 | 13 | 38
  Month 15: number analyzed (Participants) | 263 | 164 | 15 | 56
  Month 15 | 151 | 88 | 6 | 35
  Month 18: number analyzed (Participants) | 239 | 159 | 15 | 54
  Month 18 | 137 | 90 | 8 | 34
  Month 21: number analyzed (Participants) | 228 | 144 | 16 | 49
  Month 21 | 133 | 83 | 5 | 33
  Month 24: number analyzed (Participants) | 210 | 149 | 12 | 49
  Month 24 | 122 | 88 | 4 | 37

13. Secondary Outcome: Change From Baseline in DAS28-4 ESR at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated using the following formula: 0.56*square root of (TJC28) + 0.28*square root of (SJC28) + 0.70*In (ESR in mm/ hour) + 0.014*PtGA in cm. PtGA was assessed on 0-10 cm VAS scale (scores ranging from 0 cm [very well] to 10 cm [worst]), where higher scores indicated greater affliction due to disease activity). Total DAS28-4 (ESR) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity.
Time Frame: Baseline, Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Units on a scale
  Change at Month 3: number analyzed (Participants) | 399 | 253 | 55 | 79
  Change at Month 3 | -1.47 (1.49) | -1.36 (1.34) | -1.03 (1.77) | -1.69 (1.48)
  Change at Month 6: number analyzed (Participants) | 333 | 204 | 40 | 66
  Change at Month 6 | -1.52 (1.48) | -1.49 (1.41) | -0.81 (1.58) | -1.80 (1.39)
  Change at Month 9: number analyzed (Participants) | 285 | 182 | 31 | 60
  Change at Month 9 | -1.67 (1.61) | -1.56 (1.37) | -1.23 (1.66) | -1.50 (1.51)
  Change at Month 12: number analyzed (Participants) | 258 | 179 | 24 | 53
  Change at Month 12 | -1.74 (1.64) | -1.76 (1.41) | -1.81 (1.38) | -1.57 (1.49)
  Change at Month 15: number analyzed (Participants) | 226 | 152 | 13 | 49
  Change at Month 15 | -1.69 (1.54) | -1.84 (1.45) | -2.15 (0.74) | -1.70 (1.53)
  Change at Month 18: number analyzed (Participants) | 213 | 143 | 14 | 46
  Change at Month 18 | -1.63 (1.55) | -1.84 (1.44) | -2.15 (0.93) | -1.68 (1.47)
  Change at Month 21: number analyzed (Participants) | 198 | 137 | 13 | 43
  Change at Month 21 | -1.62 (1.59) | -1.72 (1.54) | -1.81 (1.32) | -1.87 (1.60)
  Change at Month 24: number analyzed (Participants) | 177 | 137 | 10 | 43
  Change at Month 24 | -1.65 (1.63) | -1.77 (1.47) | -1.85 (0.90) | -1.87 (1.51)

14. Secondary Outcome: Change From Baseline in DAS28-4 CRP at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (CRP) was calculated using the following formula: 0.56*square root of(TJC28) + 0.28*square root of(SJC28) + 0.36*ln (CRP in mg/l +1) + 0.014*(PtGA in cm)+ 0.96. PtGA was assessed on 0-10 cm VAS scale (scores ranging from 0 cm [very well] to 10 cm [worst]), where higher scores indicated greater affliction due to disease activity). Total DAS28-4 (CRP) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity.
Time Frame: Baseline, Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Units on a scale
  Change at Month 3: number analyzed (Participants) | 427 | 256 | 61 | 87
  Change at Month 3 | -1.55 (1.40) | -1.40 (1.28) | -1.04 (1.42) | -1.63 (1.35)
  Change at Month 6: number analyzed (Participants) | 347 | 210 | 46 | 73
  Change at Month 6 | -1.72 (1.43) | -1.52 (1.36) | -0.94 (1.38) | -1.90 (1.26)
  Change at Month 9: number analyzed (Participants) | 298 | 185 | 34 | 65
  Change at Month 9 | -1.82 (1.50) | -1.64 (1.22) | -1.15 (1.45) | -1.66 (1.36)
  Change at Month 12: number analyzed (Participants) | 266 | 177 | 26 | 60
  Change at Month 12 | -1.90 (1.53) | -1.79 (1.35) | -1.86 (1.32) | -1.68 (1.28)
  Change at Month 15: number analyzed (Participants) | 239 | 151 | 14 | 54
  Change at Month 15 | -1.89 (1.44) | -1.77 (1.26) | -2.13 (1.49) | -1.75 (1.39)
  Change at Month 18: number analyzed (Participants) | 212 | 140 | 14 | 52
  Change at Month 18 | -1.84 (1.49) | -1.85 (1.37) | -2.06 (1.51) | -1.62 (1.34)
  Change at Month 21: number analyzed (Participants) | 202 | 132 | 13 | 47
  Change at Month 21 | -1.81 (1.49) | -1.74 (1.47) | -1.67 (1.27) | -1.84 (1.45)
  Change at Month 24: number analyzed (Participants) | 179 | 138 | 12 | 46
  Change at Month 24 | -1.84 (1.49) | -1.79 (1.40) | -1.48 (1.04) | -1.92 (1.31)

15. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: The duration of morning stiffness was determined by asking the following questions: "When you wake up in the morning, do you currently suffer from morning stiffness?" "How long does the morning stiffness last from the time you wake up?". The change from baseline in duration of morning stiffness was calculated as: morning stiffness at time point -morning stiffness at baseline.
Time Frame: Baseline, Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Minutes
  Change at Month 3: number analyzed (Participants) | 560 | 320 | 79 | 101
  Change at Month 3 | -27.71 (86.53) | -22.23 (108.98) | -44.73 (164.97) | -26.48 (45.41)
  Change at Month 6: number analyzed (Participants) | 472 | 277 | 56 | 86
  Change at Month 6 | -29.00 (110.51) | -25.74 (126.36) | -35.18 (60.26) | -28.64 (48.50)
  Change at Month 9: number analyzed (Participants) | 411 | 235 | 46 | 78
  Change at Month 9 | -37.00 (97.53) | -36.16 (113.11) | -38.43 (70.31) | -29.55 (62.24)
  Change at Month 12: number analyzed (Participants) | 357 | 208 | 33 | 71
  Change at Month 12 | -42.11 (100.95) | -35.88 (105.09) | -27.18 (45.05) | -32.59 (57.80)
  Change at Month 15: number analyzed (Participants) | 323 | 191 | 25 | 59
  Change at Month 15 | -37.20 (123.17) | -42.20 (118.62) | -36.20 (44.26) | -35.12 (61.01)
  Change at Month 18: number analyzed (Participants) | 292 | 192 | 20 | 62
  Change at Month 18 | -41.01 (106.86) | -36.57 (107.59) | -47.95 (63.25) | -34.95 (58.77)
  Change at Month 21: number analyzed (Participants) | 270 | 161 | 15 | 52
  Change at Month 21 | -31.24 (137.43) | -28.71 (50.98) | -42.47 (58.09) | -31.13 (65.98)
  Change at Month 24: number analyzed (Participants) | 248 | 153 | 14 | 56
  Change at Month 24 | -33.12 (61.16) | -38.17 (116.88) | -26.36 (65.33) | -39.88 (61.46)

16. Secondary Outcome: Change From Baseline in the Functional Ability Questionnaire Hannover (FFbH) at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: The FFbH for RA is a German short questionnaire for the assessment of patientive functional capacity in the context of basic everyday activities (range: 0-100% functional capacity, where higher percentage indicates more capacity for everyday activities). The FFbH questionnaire consisted of 18 questions with 3 possible responses (Yes; Yes, but with effort; No or only with outside help). The total score was the sum of the scores of all 18 questions, where for each question (Yes = 2 points; Yes, but with effort = 1 point; No or only with outside help = 0 points).The functional capacity (%) is calculated by (total score*100) divided by (2*number of valid responses). The change from baseline was calculated at each time point as functional capacity at timepoint - functional capacity at baseline.
Time Frame: Baseline, Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent functional capacity
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Percent functional capacity
  Change at Month 3: number analyzed (Participants) | 578 | 328 | 83 | 103
  Change at Month 3 | 6.73 (15.08) | 5.31 (16.05) | 8.82 (15.75) | 6.52 (14.29)
  Change at Month 6: number analyzed (Participants) | 487 | 283 | 61 | 87
  Change at Month 6 | 8.73 (17.14) | 6.12 (17.23) | 10.82 (18.57) | 7.02 (15.08)
  Change at Month 9: number analyzed (Participants) | 426 | 239 | 47 | 79
  Change at Month 9 | 8.49 (16.60) | 6.45 (15.83) | 12.23 (17.22) | 5.33 (15.40)
  Change at Month 12: number analyzed (Participants) | 368 | 215 | 34 | 72
  Change at Month 12 | 8.41 (16.69) | 7.78 (17.22) | 13.59 (19.05) | 7.26 (14.58)
  Change at Month 15: number analyzed (Participants) | 337 | 195 | 24 | 60
  Change at Month 15 | 8.42 (17.64) | 8.56 (17.33) | 13.83 (19.05) | 6.55 (14.96)
  Change at Month 18: number analyzed (Participants) | 308 | 194 | 20 | 63
  Change at Month 18 | 8.20 (17.75) | 8.15 (17.42) | 17.90 (18.26) | 5.90 (14.65)
  Change at Month 21: number analyzed (Participants) | 280 | 163 | 16 | 53
  Change at Month 21 | 9.46 (19.24) | 7.43 (17.42) | 16.00 (17.36) | 4.23 (13.27)
  Change at Month 24: number analyzed (Participants) | 258 | 157 | 14 | 57
  Change at Month 24 | 9.38 (18.50) | 8.78 (17.61) | 15.21 (20.50) | 7.18 (16.00)

17. Secondary Outcome: Number of Participants Achieving Functional Remission in FFbH at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: The FFbH for RA is a German short questionnaire for the assessment of patientive functional capacity in the context of basic everyday activities (range: 0-100% functional capacity, where higher percentage indicates more capacity for everyday activities). The FFbH questionnaire consisted of 18 questions with 3 possible responses (Yes; Yes, but with effort; No or only with outside help). The total score was the sum of the scores of all 18 questions, where for each question (Yes = 2 points; Yes, but with effort = 1 point; No or only with outside help = 0 points). The functional capacity [%] is calculated by (total score*100)/ (2*number of valid responses). Functional remission in FFbH was defined as functional capacity > 83 %.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Month 3: number analyzed (Participants) | 579 | 331 | 83 | 103
  Month 3 | 174 | 114 | 18 | 47
  Month 6: number analyzed (Participants) | 489 | 285 | 62 | 88
  Month 6 | 157 | 102 | 17 | 40
  Month 9: number analyzed (Participants) | 426 | 241 | 48 | 79
  Month 9 | 139 | 84 | 14 | 34
  Month 12: number analyzed (Participants) | 369 | 217 | 34 | 72
  Month 12 | 116 | 85 | 9 | 31
  Month 15: number analyzed (Participants) | 338 | 197 | 24 | 60
  Month 15 | 122 | 84 | 6 | 25
  Month 18: number analyzed (Participants) | 309 | 196 | 20 | 63
  Month 18 | 99 | 80 | 7 | 26
  Month 21: number analyzed (Participants) | 281 | 165 | 16 | 53
  Month 21 | 99 | 65 | 7 | 19
  Month 24: number analyzed (Participants) | 258 | 159 | 14 | 57
  Month 24 | 92 | 62 | 8 | 26

18. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQoL) Group EuroQoL- 5 Dimensions- 3 Levels (EQ-5D-3L) Total Scores at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: The EQ-5D-3L is a standardised instrument used to measure quality of life. It is based on five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression with each dimension having three levels of function: 1 indicates no problem; 2 indicates some problem; 3 indicates extreme problem. Scoring formula developed by EuroQol Group (German weights) assigns a utility value for each domain in the profile. Score was transformed and results in a total score range of 0.05 to 1.00; higher scores indicating a better health state.
Time Frame: Baseline, Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Units on a scale
  Change at Month 3: number analyzed (Participants) | 573 | 324 | 82 | 101
  Change at Month 3 | 0.119 (0.205) | 0.109 (0.195) | 0.079 (0.197) | 0.102 (0.159)
  Change at Month 6: number analyzed (Participants) | 484 | 276 | 59 | 86
  Change at Month 6 | 0.134 (0.214) | 0.110 (0.217) | 0.090 (1.197) | 0.100 (0.192)
  Change at Month 9: number analyzed (Participants) | 422 | 238 | 45 | 78
  Change at Month 9 | 0.133 (0.204) | 0.118 (0.222) | 0.120 (0.188) | 0.054 (0.206)
  Change at Month 12: number analyzed (Participants) | 366 | 213 | 33 | 71
  Change at Month 12 | 0.142 (0.210) | 0.122 (0.221) | 0.087 (0.228) | 0.095 (0.173)
  Change at Month 15: number analyzed (Participants) | 336 | 194 | 23 | 59
  Change at Month 15 | 0.137 (0.223) | 0.135 (0.207) | 0.149 (0.199) | 0.102 (0.259)
  Change at Month 18: number analyzed (Participants) | 305 | 195 | 20 | 62
  Change at Month 18 | 0.140 (0.206) | 0.127 (0.209) | 0.169 (0.237) | 0.098 (0.196)
  Change at Month 21: number analyzed (Participants) | 279 | 162 | 15 | 52
  Change at Month 21 | 0.134 (0.207) | 0.122 (0.210) | 0.151 (0.202) | 0.106 (0.206)
  Change at Month 24: number analyzed (Participants) | 254 | 157 | 14 | 56
  Change at Month 24 | 0.133 (0.207) | 0.137 (0.205) | 0.163 (0.199) | 0.125 (0.226)

19. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)- Fatigue Scale at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: The FACIT-F Scale is a participant completed questionnaire consisting of 13 items that assess fatigue. Participants responded to each item on a 5-point scale based on their experience of fatigue during the past 7 days (0 = not at all; 1 = a little bit; 2 =somewhat; 3 = quite a bit; 4 = very much). Instrument scoring yielded a range from 0 to 52 (negatively worded items were reversed during analysis), with higher scores representing better participant status (less fatigue).
Time Frame: Baseline, Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Units on a scale
  Change at Month 3: number analyzed (Participants) | 568 | 323 | 80 | 98
  Change at Month 3 | 4.83 (9.63) | 3.59 (8.57) | 3.71 (9.99) | 3.35 (9.12)
  Change at Month 6: number analyzed (Participants) | 481 | 275 | 57 | 86
  Change at Month 6 | 5.57 (10.11) | 4.25 (10.11) | 5.68 (8.79) | 2.58 (9.28)
  Change at Month 9: number analyzed (Participants) | 417 | 236 | 44 | 76
  Change at Month 9 | 5.63 (9.87) | 4.44 (9.46) | 5.34 (10.93) | 1.78 (10.53)
  Change at Month 12: number analyzed (Participants) | 360 | 211 | 31 | 68
  Change at Month 12 | 5.78 (10.69) | 5.54 (9.88) | 6.61 (10.73) | 4.24 (10.49)
  Change at Month 15: number analyzed (Participants) | 331 | 193 | 21 | 58
  Change at Month 15 | 5.63 (10.57) | 5.34 (9.94) | 6.33 (12.14) | 3.31 (10.05)
  Change at Month 18: number analyzed (Participants) | 303 | 191 | 19 | 61
  Change at Month 18 | 5.96 (10.51) | 5.91 (9.92) | 13.05 (8.93) | 3.44 (8.04)
  Change at Month 21: number analyzed (Participants) | 276 | 161 | 14 | 51
  Change at Month 21 | 6.32 (11.17) | 6.65 (9.85) | 11.43 (10.62) | 4.02 (9.87)
  Change at Month 24: number analyzed (Participants) | 255 | 154 | 13 | 55
  Change at Month 24 | 6.03 (10.36) | 6.72 (9.31) | 12.69 (8.40) | 4.49 (9.68)

20. Secondary Outcome: Mean Number of Days of Drug Survival at Months 12 and 24
Description: Drug survival was assessed using Kaplan-Meier methodology. For participants who terminated tofacitinib, the drug survival status was recorded as (status = 1 and time = termination date tofacitinib - date of initiation on tofacitinib) and for participants who do not terminate tofacitinib (status = 0 and time = date of final visit - date of initiation on tofacitinib.
Time Frame: At 12 and 24 months
Population: FAS included all participants who received at least 1 dose of tofacitinib and have at least 1 set of post-baseline measurements. Here" Number Analyzed" = participants evaluable for specified rows.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Days
  Month 12: number analyzed (Participants) | 725 | 412 | 111 | 129
  Month 12 | 339.83 (5.73) | 341.17 (7.18) | 233.30 (14.00) | 337.36 (12.48)
  Month 24 | 534.49 (11.35) | 542.15 (14.28) | 317.51 (25.09) | 532.39 (25.94)

21. Secondary Outcome: Number of Participants Per Categories of Satisfaction With Tofacitinib Treatment at Months 3, 6, 9, 12, 15, 18, 21 and 24
Description: Satisfaction with treatment was assessed on a 5-point Likert scale (where 0 = extremely dissatisfied, 1= dissatisfied, 2 = neither satisfied nor dissatisfied, 3 = satisfied and 4 = extremely satisfied) in response to the question "How satisfied are you with the drugs that you have received for your arthritis since your last visit?".
Time Frame: Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
Number analyzed (Participants) | 725 | 413 | 111 | 129
Participants
  Month 3: number analyzed (Participants) | 579 | 331 | 83 | 102
  Month 3: Extremely dissatisfied | 43 | 19 | 5 | 11
  Month 3: Dissatisfied | 41 | 26 | 15 | 5
  Month 3: Neither satisfied nor dissatisfied | 107 | 63 | 22 | 20
  Month 3: Satisfied | 290 | 166 | 32 | 43
  Month 3: Extremely satisfied | 98 | 57 | 9 | 23
  Month 6: number analyzed (Participants) | 488 | 283 | 61 | 89
  Month 6: Extremely dissatisfied | 39 | 13 | 2 | 11
  Month 6: Dissatisfied | 22 | 13 | 9 | 5
  Month 6: Neither satisfied nor dissatisfied | 78 | 51 | 13 | 10
  Month 6: Satisfied | 242 | 137 | 32 | 41
  Month 6: Extremely satisfied | 107 | 69 | 5 | 22
  Month 9: number analyzed (Participants) | 422 | 240 | 48 | 80
  Month 9: Extremely dissatisfied | 27 | 11 | 0 | 4
  Month 9: Dissatisfied | 15 | 9 | 7 | 7
  Month 9: Neither satisfied nor dissatisfied | 54 | 23 | 7 | 10
  Month 9: Satisfied | 218 | 137 | 26 | 36
  Month 9: Extremely satisfied | 108 | 60 | 8 | 23
  Month 12: number analyzed (Participants) | 370 | 215 | 34 | 72
  Month 12: Extremely dissatisfied | 17 | 21 | 4 | 5
  Month 12: Dissatisfied | 14 | 5 | 0 | 1
  Month 12: Neither satisfied nor dissatisfied | 38 | 21 | 7 | 11
  Month 12: Satisfied | 207 | 117 | 19 | 38
  Month 12: Extremely satisfied | 94 | 51 | 4 | 17
  Month 15: number analyzed (Participants) | 336 | 197 | 25 | 60
  Month 15: Extremely dissatisfied | 16 | 10 | 0 | 4
  Month 15: Dissatisfied | 15 | 6 | 1 | 0
  Month 15: Neither satisfied nor dissatisfied | 37 | 24 | 5 | 8
  Month 15: Satisfied | 170 | 105 | 13 | 26
  Month 15: Extremely satisfied | 98 | 52 | 6 | 22
  Month 18: number analyzed (Participants) | 308 | 194 | 20 | 63
  Month 18: Extremely dissatisfied | 14 | 11 | 0 | 2
  Month 18: Dissatisfied | 12 | 5 | 1 | 2
  Month 18: Neither satisfied nor dissatisfied | 32 | 17 | 0 | 7
  Month 18: Satisfied | 156 | 107 | 12 | 29
  Month 18: Extremely satisfied | 94 | 54 | 7 | 23
  Month 21: number analyzed (Participants) | 277 | 163 | 15 | 53
  Month 21: Extremely dissatisfied | 12 | 9 | 0 | 4
  Month 21: Dissatisfied | 11 | 4 | 1 | 1
  Month 21: Neither satisfied nor dissatisfied | 20 | 15 | 0 | 2
  Month 21: Satisfied | 137 | 88 | 9 | 29
  Month 21: Extremely satisfied | 97 | 47 | 5 | 17
  Month 24: number analyzed (Participants) | 257 | 158 | 14 | 57
  Month 24: Extremely dissatisfied | 17 | 13 | 2 | 6
  Month 24: Dissatisfied | 5 | 2 | 1 | 0
  Month 24: Neither satisfied nor dissatisfied | 19 | 16 | 3 | 3
  Month 24: Satisfied | 135 | 73 | 5 | 26
  Month 24: Extremely satisfied | 81 | 54 | 3 | 22

ADVERSE EVENTS:
Time Frame: From date of first prescription of tofacitinib up to 24 months (maximum up to 24 Months)
Description: The safety analysis set included all participants who had received at least one dose of tofacitinib.
Arm/Group | Tofacitinib Monotherapy | Tofacitinib+Methotrexate (MTX) Combination Therapy | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy
All-Cause Mortality (participants affected / at risk) | 6/779 | 5/440 | 0/111 | 0/129
Serious Adverse Events (participants affected / at risk) | 141/779 | 69/440 | 24/111 | 27/129
Other Adverse Events (participants affected / at risk) | 402/779 | 240/440 | 81/111 | 84/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib Monotherapy (N=779) | Tofacitinib+Methotrexate (MTX) Combination Therapy (N=440) | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy (N=111) | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy (N=129)
Drug ineffective (General disorders) | 13 | 9 | 6 | 3
Therapeutic product effect incomplete (General disorders) | 7 | 3 | 2 | 3
Therapeutic product effect decreased (General disorders) | 5 | 1 | 3 | 0
Drug intolerance (General disorders) | 2 | 2 | 0 | 2
Death (General disorders) | 1 | 2 | 0 | 0
Pain (General disorders) | 1 | 2 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0 | 1
Condition aggravated (General disorders) | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Withdrawal syndrome (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 6 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 3 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 1 | 2 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 2 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1
Whipple's disease (Infections and infestations) | 1 | 0 | 0 | 1
Abscess oral (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis E (Infections and infestations) | 0 | 1 | 0 | 0
Herpes pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 0
Medical device site infection (Infections and infestations) | 0 | 1 | 0 | 0
Medical device site joint infection (Infections and infestations) | 1 | 0 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 | 4 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Carpal collapse (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 8 | 1 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 1
Aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Essential hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 4 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Medication error (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Product dose omission issue (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Vulval cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colon operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0
Osteotomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Pulmonary resection (Surgical and medical procedures) | 0 | 1 | 0 | 0
Spinal fusion surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0
Spinal operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Tenoplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Paraesthesia ear (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lipoedema (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Corneal oedema (Eye disorders) | 0 | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Contrast media reaction (Immune system disorders) | 0 | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib Monotherapy (N=779) | Tofacitinib+Methotrexate (MTX) Combination Therapy (N=440) | Tofacitinib Monotherapy To Tofacitinib+ MTX Combination Therapy (N=111) | Tofacitinib+ MTX Combination Therapy to Tofacitinib Monotherapy (N=129)
Drug ineffective (General disorders) | 69 | 42 | 11 | 15
Therapeutic product effect decreased (General disorders) | 36 | 21 | 12 | 9
Influenza like illness (General disorders) | 26 | 21 | 7 | 3
Therapeutic product effect incomplete (General disorders) | 21 | 15 | 14 | 5
Fatigue (General disorders) | 11 | 7 | 1 | 2
Oedema peripheral (General disorders) | 6 | 2 | 0 | 1
Condition aggravated (General disorders) | 1 | 3 | 1 | 0
Drug intolerance (General disorders) | 1 | 1 | 1 | 2
Pain (General disorders) | 2 | 0 | 2 | 0
Chills (General disorders) | 0 | 3 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0
Cyst (General disorders) | 2 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 1
Oedema (General disorders) | 2 | 0 | 0 | 0
Peripheral swelling (General disorders) | 2 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Drug tolerance decreased (General disorders) | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Remission not achieved (General disorders) | 0 | 1 | 0 | 0
Sense of oppression (General disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 10 | 17 | 3 | 4
Herpes zoster (Infections and infestations) | 18 | 8 | 2 | 5
Respiratory tract infection (Infections and infestations) | 17 | 11 | 2 | 1
Bronchitis (Infections and infestations) | 14 | 5 | 3 | 2
Urinary tract infection (Infections and infestations) | 11 | 6 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 8 | 2 | 1
COVID-19 (Infections and infestations) | 5 | 6 | 2 | 0
Gastrointestinal infection (Infections and infestations) | 2 | 4 | 2 | 0
Oral herpes (Infections and infestations) | 2 | 5 | 0 | 1
Conjunctivitis (Infections and infestations) | 2 | 2 | 0 | 1
Coronavirus infection (Infections and infestations) | 3 | 2 | 0 | 0
Herpes simplex (Infections and infestations) | 3 | 2 | 0 | 0
Infection (Infections and infestations) | 4 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 0 | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 2 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 2 | 0 | 0
Febrile infection (Infections and infestations) | 2 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 1 | 0 | 0
Root canal infection (Infections and infestations) | 3 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 2 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 1 | 1 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 1 | 0 | 0
Infection susceptibility increased (Infections and infestations) | 1 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 2 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Borrelia infection (Infections and infestations) | 0 | 0 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0
Infected bite (Infections and infestations) | 1 | 0 | 0 | 0
Nasal herpes (Infections and infestations) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Rotavirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 19 | 12 | 6 | 10
Diarrhoea (Gastrointestinal disorders) | 10 | 13 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 9 | 5 | 2 | 2
Vomiting (Gastrointestinal disorders) | 4 | 3 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 5 | 3 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 5 | 3 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 4 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 1 | 0
Gastritis (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Oral mucosa erosion (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Coating in mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatic failure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Regurgitation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 11 | 10 | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal instability (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 24 | 7 | 6 | 2
Dizziness (Nervous system disorders) | 12 | 16 | 4 | 1
Sciatica (Nervous system disorders) | 1 | 3 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 2 | 0 | 1
Dizziness postural (Nervous system disorders) | 2 | 0 | 0 | 0
Migraine (Nervous system disorders) | 2 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0
Hypokinesia (Nervous system disorders) | 1 | 0 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0 | 0
Movement disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Pseudoradicular syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 5 | 3 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculovesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Weight increased (Investigations) | 9 | 1 | 1 | 2
Hepatic enzyme increased (Investigations) | 2 | 4 | 2 | 1
Weight decreased (Investigations) | 1 | 2 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0
Blood glucose increased (Investigations) | 2 | 0 | 0 | 0
Borrelia test positive (Investigations) | 0 | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase abnormal (Investigations) | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 1 | 0 | 0 | 0
Lung diffusion test decreased (Investigations) | 0 | 0 | 0 | 1
Lymphocyte morphology abnormal (Investigations) | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 1 | 0
Platelet count abnormal (Investigations) | 0 | 0 | 1 | 0
Pulmonary function test decreased (Investigations) | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 1
Transaminases abnormal (Investigations) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 7 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 4 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Intentional dose omission (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Adverse event following immunisation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Mallet finger (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Palate injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Product administration error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 3 | 2 | 1
Lymphoedema (Vascular disorders) | 2 | 2 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 1 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 1 | 0
Essential hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0
Vascular pain (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Lipid metabolism disorder (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Lipoedema (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 6 | 2 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 3 | 0 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Listless (Psychiatric disorders) | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Panic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 4 | 2 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 2 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Bladder discomfort (Renal and urinary disorders) | 0 | 1 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 3 | 1 | 1 | 1
Glaucoma (Eye disorders) | 3 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Episcleritis (Eye disorders) | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0
Eyelid thickening (Eye disorders) | 1 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0
Periorbital swelling (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Bone marrow oedema (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 4 | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 2 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Eustachian tube disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Fatty liver alcoholic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 1 | 1 | 0
Thyroid disorder (Endocrine disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1
Shoulder operation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 2 | 1 | 1 | 0
Synoviorthesis (Surgical and medical procedures) | 1 | 0 | 0 | 0
Sensation of oppression (General disorders) | 0 | 1 | 0 | 0
Joint surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0
Formication (Nervous system disorders) | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03387423/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT03387423/SAP_001.pdf